CLINICAL TRIAL: NCT00600496
Title: A Phase I, Open-Label, Multi-center Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD6244 (ARRY-142886) When Given in Combination With Standard Doses of Selected Chemotherapies to Patients With Advanced Solid Tumors
Brief Title: A Phase I, Open-Label, Multi-center Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD6244 (ARRY-142886)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1532C00004
Record Dates: First submitted 2008-01-15; First posted 2008-01-25 (Estimated); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Breast Neoplasms; Colon Cancer; Colonic Cancer; Colon Neoplasms; Lung Cancer; Melanoma; Kidney Cancer
Keywords: ARRY-142886; AZD6244; Cancer; Colon Cancer; Breast Cancer; Lung Cancer; Melanoma; Kidney Cancer
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Lung Neoplasms; Melanoma; Kidney Neoplasms; Neoplasms | interventions — AZD 6244; Dacarbazine; Erlotinib Hydrochloride; Docetaxel; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): AZD6244 + docetaxel
  Interventions: Drug: AZD6244; Drug: Docetaxel
- 2 (Experimental): AZD6244 + Dacarbazine
  Interventions: Drug: AZD6244; Drug: Dacarbazine
- 3 (Experimental): AZD6244 + Erlotinib
  Interventions: Drug: AZD6244; Drug: Erlotinib
- 4 (Experimental): AZD6244 + Temsirolimus
  Interventions: Drug: AZD6244; Drug: Temsirolimus

INTERVENTIONS:
Drug: AZD6244 — twice daily oral dose
  Other Names: ARRY-142886
Drug: Dacarbazine — intravenous infusion
  Arms: 2
Drug: Erlotinib — daily oral dose
  Arms: 3
Drug: Docetaxel — intravenous infusion
  Other Names: Taxotere®
  Arms: 1
Drug: Temsirolimus — intravenous infusion
  Arms: 4

SUMMARY:
This study is being conducted to determine if a combination of AZD6244 given orally twice a day with standard doses of selected chemotherapies will be safe and tolerable for cancer patients with advanced solid tumors. The highest tolerated dose of AZD6244 in combination with selected chemotherapies will be evaluated. The study will also investigate how AZD6244 in combination with standard chemotherapies are absorbed, distributed and excreted by the body as well as the length of time that the drugs remain in the body. Initial and periodic assessments will establish patient response to the combination therapies

ELIGIBILITY:
Inclusion Criteria:

* Patients will have measurable and/or non-measurable disease, lacking curative options for whom the selected chemotherapy agents represent the standard of care
* WHO performance status 0-1
* Patients must be able to swallow AZD6244 capsules

Exclusion Criteria:

* Prior treatment with a MEK inhibitor
* Participation in a clinical study during the last 30 days or have not recovered from side effects of an investigational study drug
* Brain metastases or spinal cord compression unless treated and stable (for at least 1 month) off steroids

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-12-14 (Actual); Primary Completion 2010-08-20 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of twice daily oral doses of AZD6244 when administered in combination with standard doses of selected chemotherapies. | 28 days +
  Incidence and intensity of adverse events as graded by CTCAE (version 3.0), physical examinations, vital signs (including weight, blood pressure and pulse rate), ECG parameters, MUGA scan and echocardiography, clinical chemistry (including liver function tests), Brain Natriuretic Peptide (BNP), Troponin I, hematology, urinalysis, and ophthalmologic examinations.

SECONDARY OUTCOMES:
PK of AZD6244 and selected chemotherapies. | Cycle 1 Day 3 and Cycle 2 day 1
  The PK parameters will be derived using noncompartmental analysis. The maximum plasma concentrations (Cmax) and the time to reach the maximum plasma concentrations (tmax) will be determined by visual inspection of the plasma concentration-time profiles. The area under the plasma concentration-time curve from zero to 12 hours post dose, AUC(0-12), will be calculated by the linear trapezoidal rule. Where more than one maxima occurs, the reported value will be assigned to the first occurrence.
Define highest tolerated dose of AZD6244 when in combination with selected chemotherapies. | 28 days +
  The starting dose of AZD6244 in each arm will be 50mg. Continuous dosing (commencing Cycle 1/Day 3 for docetaxel and dacarbazine and Cycle 1/Day 8 for erlotinib and temsirolimus) will be BD. The AZD6244 dose may be maintained or reduced.
Tumor response. | 28 days +
  To make a preliminary assessment of tumor response as measured by Objective Response Rate (ORR) per investigator's assessment using Response Evaluation Criteria in Solid Tumors (RECIST) when AZD6244 Hyd-Sulfate is given in combination with standard doses of selected chemotherapies.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia LoRusso, DO, Principal Investigator — Barbara Ann Karmanos Cancer Institute; Roger Cohen, MD, Principal Investigator — Fox Chase Cancer Center; Jeffrey Infante, MD, Principal Investigator — SCRI Development Innovations, LLC; Kevin Kim, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Research Site, Detroit, Michigan
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Infante JR, Cohen RB, Kim KB, Burris HA 3rd, Curt G, Emeribe U, Clemett D, Tomkinson HK, LoRusso PM. A phase I dose-escalation study of Selumetinib in combination with Erlotinib or Temsirolimus in patients with advanced solid tumors. Invest New Drugs. 2017 Oct;35(5):576-588. doi: 10.1007/s10637-017-0459-7. Epub 2017 Apr 19. PMID 28424891
- [Derived] LoRusso PM, Infante JR, Kim KB, Burris HA 3rd, Curt G, Emeribe U, Clemett D, Tomkinson HK, Cohen RB. A phase I dose-escalation study of selumetinib in combination with docetaxel or dacarbazine in patients with advanced solid tumors. BMC Cancer. 2017 Mar 6;17(1):173. doi: 10.1186/s12885-017-3143-6. PMID 28264648
- [Derived] Patel SP, Lazar AJ, Papadopoulos NE, Liu P, Infante JR, Glass MR, Vaughn CS, LoRusso PM, Cohen RB, Davies MA, Kim KB. Clinical responses to selumetinib (AZD6244; ARRY-142886)-based combination therapy stratified by gene mutations in patients with metastatic melanoma. Cancer. 2013 Feb 15;119(4):799-805. doi: 10.1002/cncr.27790. Epub 2012 Sep 12. PMID 22972589
- See also: D1532C00004 Clinical Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1170&filename=D1532C00004_Study_Synopsis.pdf